CLINICAL TRIAL: NCT02724904
Title: A Pilot Study of Reduced Intensity Conditioning Allogeneic Hematopoietic Stem Cell Transplantation for Patients With Relapsed CNS Involvement by Lymphoma
Brief Title: Reduced Intensity Conditioning Allogeneic Hematopoietic Stem Cell Transplant (HSCT) For Lymphoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Drug logistics
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Adienne SA (Industry); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Yi-Bin A. Chen, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-433
Record Dates: First submitted 2016-01-14; First posted 2016-03-31 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Lymphoma
Keywords: Allogeneic hematopoietic stem cell transplantation; CNS Non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Bone Marrow Transplantation; fludarabine; fludarabine phosphate; Thiotepa; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Allogeneic Stem Cell Transplantation (Experimental): Patients will undergo reduced intensity conditioning (fludarabine and thiotepa) followed by fully matched related or unrelated allogeneic stem cell transplantation. Afterwards, patients will receive standard post-transplant care (Methotrexate).
  Interventions: Procedure: Allogeneic stem cell transplantation; Drug: Fludarabine; Drug: Thiotepa; Drug: Methotrexate

INTERVENTIONS:
Procedure: Allogeneic stem cell transplantation — Reduced intensity allogeneic stem cell transplantation from a fully matched related or unrelated donor
  Other Names: bone marrow transplant
Drug: Fludarabine — Standard Treatment
  Other Names: Fludara
Drug: Thiotepa — Standard Treatment
  Other Names: Thioplex
Drug: Methotrexate — IV Bolus
  Other Names: Otrexup™

SUMMARY:
This research study is assessing the feasibility of reduced intensity allogeneic hematopoietic stem cell transplantation (HSCT) as a possible treatment for relapsed / refractory non-Hodgkin lymphoma involving the central nervous system (CNS). HSCT is the transplantation of stem cells, usually derived from bone marrow, peripheral blood, or umbilical cord blood.

DETAILED DESCRIPTION:
This research study is a Pilot Study, which is the first time investigators are examining this study intervention (allogeneic stem cell transplantation) for this population (patients with CNS lymphoma), which is a type of stem cell transplantation.

Historically, patients with central nervous system (CNS) involvement by non-Hodgkin lymphoma (NHL) have had high rates of disease relapse after initial therapy. Given these poor outcomes with conventional chemotherapy, more intense treatment with high-dose chemotherapy and autologous stem cell transplantation (ASCT) has been explored, yet relapse remains an issue. For older patients, ASCT may not be feasible given the inability to tolerate high-doses of chemotherapy.

In patients with systemic NHL who relapse after ASCT or cannot tolerate ASCT, yet are responsive to chemotherapy, allogeneic stem cell transplant is often considered. Allogeneic transplantation is thought to work by giving the recipient an entirely new blood system from a donor. This new blood system includes a new immune system which can hopefully attack any lymphoma much like it would attack a bacterial or viral infection. Currently, this is one established standard of care for patients with lymphoma of the body who relapse after initial chemotherapy treatment. The investigators are testing if this treatment can be extended to patients with lymphoma of the central nervous system.

The following chemotherapy drugs included in this study which will be administered: Fludarabine, Thiotepa, and Methotrexate. The FDA (the U.S. Food and Drug Administration) has approved these chemotherapy agents individually as a treatment option for your disease. The combination has not been approved by the FDA. Thiotepa and Methotrexate have been shown to pass through the blood-brain barrier, a highly selective barrier that restricts many chemicals from entering the brain and spinal cord. Fludarabine is the backbone chemotherapy in all reduced intensity conditioning regimens.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed non-Hodgkin lymphoma involving the central nervous system (CNS) as defined by:

  * Biopsy of CNS mass in the brain, parenchyma, leptomeninges, or spinal cord demonstrating NHL.
  * Ocular biopsy from retina, subretinal pigment epithelial space, or optic nerve, or vitrectomy specimen, demonstrating NHL.
  * Biopsy of mass lesion outside of the CNS, or blood or body fluid specimen, documenting NHL, in conjunction with brain or spinal CT, PET/CT (positron emission tomography / computed tomography), or MRI showing radiographic abnormalities characteristic of CNS involvement with lymphoma.
  * CSF cytology demonstrating a malignant clonal NHL population, consistent with lymphomatous leptomeningitis, with or without a radiographically or pathologically identifiable CNS or systemic mass lesion. Patients with CSF (cerebral spinal fluid) studies negative for NHL by cytology but positive for a monoclonal population by flow cytometry and/or molecular PCR (polymerase chain reaction) studies may be eligible if they have radiographic evidence of a CNS lymphoma or if they have symptoms clinically consistent with CNS lymphomatous involvement; for such cases, please contact the protocol chair, Dr. Yi Bin Chen, to discuss eligibility prior to enrollment.
* Patients must have experienced relapsed disease after high-dose chemotherapy with autologous stem cell transplantation (ASCT) OR have experienced relapse / progression on first-line high-dose methotrexate-based therapy and are not candidates for ASCT in the judgment of the treating physician. Discussion with the PI is encouraged for the latter scenario.
* All participants must demonstrate a partial or complete response (PR or CR) of their CNS and systemic disease to pre-enrollment therapy and must be in PR or CR at the time of enrollment. Acceptable therapies include systemic or intrathecal chemo/immunotherapy and/or radiotherapy as well as corticosteroids.
* Age ≥ 18 years as this study will be open at sites which treat adults.
* ECOG (Eastern Cooperative Oncology Group) performance status ≤ 2 (Karnofsky score ≥ 60%, see Appendix A).
* Participants must have adequate organ function as defined below:

  * Total serum bilirubin within normal institutional limits (unless patient has Gilbert's syndrome, where then direct serum bilirubin should be within normal institutional limits).
  * AST (SGOT) / ALT(SGPT) ≤ 3× institutional upper limit of normal.
  * Serum creatinine within normal institutional limits

    --- OR
  * Creatinine clearance ≥ 50 mL/min/1.73 m2 for participants with creatinine level above institutional normal.
  * Left ventricular ejection fraction ≥ 40% measured either by echocardiogram or nuclear cardiac scan.
  * FEV1 (forced expiratory volume in 1 second), FVC (forced vital capacity) and DLCO all ≥ 50% of predicted (DLCO corrected for hemoglobin).
* Participants must have a well-matched adult donor willing to donate peripheral blood stem cells with well-matched defined as: 8/8 matched related or unrelated donor (HLA-A, B, C, DRB1 by allele level).
* Because chemotherapy agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 12 months after the date of stem cell transplantation.
* Ability to understand and the willingness to sign a written informed consent document.
* Eligibility Criteria for Donors

  * Donors must be medically fit to donate peripheral blood stem cells through standard G-CSF mobilization as assessed by institutional or unrelated marrow registry standards.
  * Donors will not have to sign a study specific informed consent to participate given that donors will be undergoing standard G-CSF mobilization and leukapheresis.
* Exclusion Criteria:
* Participants who have had chemotherapy or radiotherapy within 4 weeks prior to the 1st day of conditioning chemotherapy.
* Participants who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to fludarabine, thiotepa or other agents used in study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or lactating women are excluded from this study because they are routinely ineligible to be treated with allogeneic stem cell transplantation.
* HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for increased risk of lethal infections when treated with marrow-suppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Treatment-related mortality (TRM) | From date of transplant to 6 months afterwards
  Death from a non-relapse cause

SECONDARY OUTCOMES:
Percentage of Participants that experienced grade II-IV acute graft-vs-host disease (GVHD) | From date of transplant to 6 months afterwards
  Cumulative incidence of acute GVHD
Progression-free survival (PFS) | From date of transplant to disease progression or death, whichever occurred first, and patients who are alive without disease progression will be censored at last day known alive in the first 2 years after transplant
  Relapse or death
Overall survival (OS) | From time of transplant to death, or last day known alive in the first 2 years after transplant
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Bin Chen, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No